CLINICAL TRIAL: NCT02090777
Title: Health Coaching for Glaucoma Patients, Pilot Study
Brief Title: Health Coaching for Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00052498
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-01

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Health Coach (Other): Health Coach is conducted to see if it improves ophthalmic care for glaucoma patients.
  Interventions: Behavioral: Health Coach

INTERVENTIONS:
Behavioral: Health Coach

SUMMARY:
The study will be conducted to examine the feasibility of using a Health Coach for improving the ophthalmic care of glaucoma patients. Patients taking glaucoma medications will have a coaching intervention and adherence to glaucoma drops will be monitored using a dose-recording device. The dosing data will be analyzed to examine the effect on adherence and qualitative interviews at the conclusion of the study will be used to examine which elements of the coaching experience were most helpful in the glaucoma patient population.

DETAILED DESCRIPTION:
Glaucoma medication adherence will be tracked using a dose recording device to record eye drop usage.

ELIGIBILITY:
Inclusion Criteria:

* Adult whose age is >18 years
* Diagnosed with glaucoma
* Patient of Duke Glaucoma Service
* Prescribed or using topical glaucoma eye medication for at least 6 months
* Primarily self-administering his or her eye drops
* English speaking
* Patient should be able to use the telephone for the coaching intervention,
* Patient should be available by phone to complete the coaching intervention
* Patient should be willing and able to use the MEMS (Medication Event Monitoring System) device for recording medication use
* Patient must be willing and able to come to the Eye Center for an exit interview and to return the MEMS device
* Patient must be able to give consent

Exclusion Criteria:

* Patient should be excluded if he or she may need glaucoma surgery or laser during the 6 months of the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jullia Rosdahl, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 participants signed consent. 5 participants decided not to participate after signing consent and did not start study. 4 participants started and completed the study.
Groups:
- Health Coach: Health Coach is conducted to see if it improves ophthalmic care for glaucoma patients.
  Health Coach
Period: Overall Study
Arm/Group | Health Coach
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed this pilot study intervention are included in the analysis.
Arm/Group | Health Coach
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 73 [69 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Glaucoma Medication Adherence
Description: Glaucoma medication adherence will be tracked using a dose recording device to record eye drop usage. The average of the participants percentage of time they adhered to using the medication will be reported.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: percentage of adherence time
Arm/Group | Health Coach
Number analyzed (Participants) | 4
percentage of adherence time | 72 (27)

ADVERSE EVENTS:
Arm/Group | Health Coach
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No